CLINICAL TRIAL: NCT03967990
Title: Evaluating the Effects of Corn Flour Consumption on Cardio-metabolic Outcomes and the Gut Microbiome in Adults With High Cholesterol
Brief Title: Corn and Heart Health Study
Acronym: CHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: North American Millers Association - Corn Division (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00007518
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Gut Microbiome; Cholesterol, LDL; Cholesterol, HDL
Keywords: cholesterol; gut microbiome; gut microbiota; dietary fiber; whole grain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- refined-50/50-whole (Experimental): 48 g/d of corn flour was delivered to participants in two daily 24 g servings as pita breads and/or muffins via (1) refined cornmeal flour, followed by (2) 50/50 mix of refined cornmeal flour plus corn bran, followed by (3) whole grain cornmeal flour
  Interventions: Other: Refined cornmeal flour; Other: 50/50 refined cornmeal-bran mix; Other: Whole grain cornmeal flour
- 50/50-whole-refined (Experimental): 48 g/d of corn flour was delivered to participants in two daily 24 g servings as pita breads and/or muffins via (1) 50/50 mix of refined cornmeal flour plus corn bran, followed by (2) whole grain cornmeal flour, followed by (3) refined cornmeal flour
  Interventions: Other: Refined cornmeal flour; Other: 50/50 refined cornmeal-bran mix; Other: Whole grain cornmeal flour
- whole-refined-50/50 (Experimental): 48 g/d of corn flour was delivered to participants in two daily 24 g servings as pita breads and/or muffins via (1) whole grain cornmeal flour, followed by (2) refined cornmeal flour, followed by (3) 50/50 mix of refined cornmeal flour plus corn bran
  Interventions: Other: Refined cornmeal flour; Other: 50/50 refined cornmeal-bran mix; Other: Whole grain cornmeal flour
- refined-whole-50/50 (Experimental): 48 g/d of corn flour was delivered to participants in two daily 24 g servings as pita breads and/or muffins via (1) refined cornmeal flour, followed by (2) whole grain cornmeal flour, followed by (3) 50/50 mix of refined cornmeal flour plus corn bran
  Interventions: Other: Refined cornmeal flour; Other: 50/50 refined cornmeal-bran mix; Other: Whole grain cornmeal flour
- 50/50-refined-whole (Experimental): 48 g/d of corn flour was delivered to participants in two daily 24 g servings as pita breads and/or muffins via (1) 50/50 mix of refined cornmeal flour plus corn bran, followed by (2) refined cornmeal flour, followed by (3) whole grain cornmeal flour
  Interventions: Other: Refined cornmeal flour; Other: 50/50 refined cornmeal-bran mix; Other: Whole grain cornmeal flour
- whole-50/50-refined (Experimental): 48 g/d of corn flour was delivered to participants in two daily 24 g servings as pita breads and/or muffins via (1) whole grain cornmeal flour, followed by (2) 50/50 mix of refined cornmeal flour plus corn bran, followed by (3) refined cornmeal flour
  Interventions: Other: Refined cornmeal flour; Other: 50/50 refined cornmeal-bran mix; Other: Whole grain cornmeal flour

INTERVENTIONS:
Other: Refined cornmeal flour — 48 g/d of refined cornmeal flour served to participants as two daily 24 g servings via pita breads and/or muffins
Other: 50/50 refined cornmeal-bran mix — 48 g/d of a mix of 50% refined cornmeal flour and 50% corn bran flour served to participants as two daily 24 g servings via pita breads and/or muffins
Other: Whole grain cornmeal flour — 48 g/d of whole grain cornmeal flour served to participants as two daily 24 g servings via pita breads and/or muffins

SUMMARY:
The purpose of this study is to investigate the effects of 3 different corn flours: (1) whole grain corn flour, (2) 50% refined corn flour + 50% corn bran derived from whole corn meal, and (3) refined corn flour, on cardio-metabolic outcomes and changes in the gut microbiome.

DETAILED DESCRIPTION:
Dietary fibers are extremely complex and foster health in a variety of ways that are not fully understood. The Adequate Intake of fiber (14 g per 1000 kcal consumed) is based on data that strongly support a relationship with cardiovascular disease prevention (Slavin, 2013). While cereal fibers have been shown to be most effective at reducing cardiovascular disease risk (IOM, 2002), the components of dietary fiber (e.g. germ, bran) that exert this effect remain inadequately studied in cardiometabolic outcomes. Further, specific types of dietary fiber (natural and synthetic) have been shown to increase beneficial microbial species in the gastrointestinal tract, which are accompanied by improvements in inflammatory and metabolic disease markers. Very little is known about how isolated or intact fiber in whole grains solicit beneficial health effects via microbial mechanisms. Our goal is to study both changes in cardiometabolic outcomes and the gut microbiome after consuming different types of corn-based meals.

Aim 1: To evaluate cardio-metabolic outcomes (primary outcome: LDL cholesterol) after consuming 48 g/d of whole grain corn flour, 50% refined corn flour + 50% corn bran derived from whole corn meal, and refined corn flour for 4 weeks in adult males and females with elevated LDL cholesterol in a crossover design.

Aim 2: To evaluate changes in the gut microbiome after consuming 48 g/d of whole grain corn flour, 50% refined corn flour + 50% corn bran derived from whole corn meal, and refined corn flour for 4 weeks in adult males and females with elevated LDL cholesterol in a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy English and Spanish speaking males and females with elevated circulating cholesterol levels (LDL-c ≥ 120 mg/dL).
* Individuals with LDL-c > 190 mg/dL will be permitted to participate but must provide a letter from their doctor stating that they are comfortable with their participation in the study.

Exclusion Criteria:

* recent weight fluctuations (> 5 lb in past 3 months), following specialized or restrictive diets (e.g. carbohydrate restriction, veganism)
* use of supplements (antioxidants, fiber, botanicals)
* allergies to dairy, egg, wheat, corn or gluten
* use of antibiotics in the past 2-3 months
* use of lipid lowering medications
* regular physical activity ≥ 30 min/d for ≥ 5 days/wk
* history of thyroid disorders, diabetes, heart disease, cancer, hepatitis, inflammatory conditions and/or gastrointestinal disorders which may impact gut function and metabolism
* anyone with a fear of needles or blood draws
* If female, women may not be pregnant or lactating during the study.
* Unwillingness to comply with study protocols will also result in exclusion from the study.
* Participants in this study will not be eligible if they are participating in other research studies at the same time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
LDL Cholesterol | 0 weeks, 4 weeks
  Serum LDL cholesterol concentrations will be measured at the 0 and 4 weeks for each cornmeal intervention
HDL Cholesterol | 0 weeks, 4 weeks
  Serum HDL cholesterol concentrations will be measured at the 0 and 4 weeks for each cornmeal intervention

SECONDARY OUTCOMES:
Gut Microbiome Diversity | 0 weeks, 4 weeks
  Fecal gut microbiome communities will be sequenced using microbial DNA extracted from samples at 0 and 4 weeks for each cornmeal intervention. Amplified copies of the 16S rRNA gene will be evaluated for treatment differences in alpha (within-sample richness and evenness) and beta diversity (between-sample community structure). Relative and differential abundance of individual microbial taxa will also be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Corrie M Whisner, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liedike B, Khatib M, Tabarsi B, Harris M, Wilson SL, Ortega-Santos CP, Mohr AE, Vega-Lopez S, Whisner CM. Evaluating the Effects of Corn Flour Product Consumption on Cardiometabolic Outcomes and the Gut Microbiota in Adults with Elevated Cholesterol: A Randomized Crossover. J Nutr. 2024 Aug;154(8):2437-2447. doi: 10.1016/j.tjnut.2024.06.003. Epub 2024 Jun 14. PMID 38880174